CLINICAL TRIAL: NCT03212079
Title: Novel Individualized Intervention for Behavioral Change Among High-Risk Group Cancer Survivors : Physical Activities by Technology Help (PATH)
Brief Title: Physical Activities by Technology Help (PATH)
Acronym: PATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00113882
Record Dates: First submitted 2017-04-04; First posted 2017-07-11 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer; Prostate Cancer; Lung Cancer; Colorectal Cancer; Cervical Cancer; Oral Cancer
Keywords: Cancer Survivors; Physical Activities; Baltimore; State of Maryland
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Uterine Cervical Neoplasms; Mouth Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: This is a single center three arms randomized trial.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): The participant will self motivate hi/herself to increase physical activities.
- Mycoach Smart Text (Experimental): The participant will receive personalized smart text messages to encourage him/her to increase physical activities
  Interventions: Behavioral: Mycoach Smart Text
- MyCoach via Amazon Alexa (Experimental): The participant will interact with intelligent coach on Amazon Alexa (a digital voice assist) to help him/her become more active
  Interventions: Behavioral: MyCoach on Amazon Alexa

INTERVENTIONS:
Behavioral: Mycoach Smart Text — Personalized text messages to you cellphone to help you become more active
  Other Names: Smart text
  Arms: Mycoach Smart Text
Behavioral: MyCoach on Amazon Alexa — This is an intelligent voice that you can communicate with via Amazon echo speaker
  Other Names: Digital Voice Assist
  Arms: MyCoach via Amazon Alexa

SUMMARY:
PATH is a research study for cancer survivors to help participants to become more active. Studies suggested an association between inactivity and cancer. The investigators created new novel ways and technologies that may help participants to become more active. The three methods the investigators are studying are: 1) participant become active on her/his own; educational material will be provided; 2) working with a programmed health coach over the phone via text messages; and 3) using digital voice assist to help participant become more active. The digital voice assist will be delivered via Amazon Alexa on Echo speaker (it is the famous intelligent voice that you see in superball commercial by Alec Baldwin). This study is funded by the State of Maryland.

DETAILED DESCRIPTION:
If the participant agree to be in this study, the investigators will ask the participant to do the following things:

The participant will be asked questions about his/her physical activity (walking, running or other exercise) to determine if he/she are eligible to participate. If the participant is eligible and interested in participating, the investigators will ask hi/her to read and sign the consent form.

After that, the investigators will randomly assign the participant to a research group (this method would be similar to drawing numbers from a hat). The result will determine which group the participant will belong to. The study would have three different groups:

1. Group one will be self-motivated to be physically active (control group)
2. The second group will receive smart daily text messages only (text group);
3. The last group would have the Amazon Echo smart device installed in participants' homes and they will interact with a digital voice assist that will help them be active (Alexa group).

   * All study participants will receive a Fitbit device which you can keep after the study.
   * When the investigators start the study, the participant will be asked to start wearing wrist device immediately. For the next one week the investigators will monitor the participant daily number of steps to establish how active he/she is. The participant will not be required to change his/her daily routine in the first week.
   * After the end of the first week, the investigators will ask the participant to increase his/her daily steps to at least 10 thousand steps per day for the next four weeks. In total the participant will have one week of hi/her normal daily routine and four weeks of trying to do 10 thousand steps per day or more.
   * If the participant is in the control group, the investigators will ask you to try to do 10 thousand steps per day on his/her own.
   * If the participant are in the text group, he/she will get smart text messages with healthy tips to help track his/her activities and reach his/her daily goal.
   * If the participant is in Alexa group, a study member will visit the participant at his/her home before the end of the first week to install the Echo smart speaker and to explain to the participant how to use the voice assist to help him/her become more active for the next four weeks.

ELIGIBILITY:
Inclusion Criteria:

* A cancer survivor of breast, prostate, lung, colorectal, cervical or oral cancer survivor and live within the Baltimore Maryland area.
* Finished your active cancer treatment at least three months ago.
* Overweight or obese and do not exercise daily.
* Do not have any physical limitation to do mild to moderate physical activities.
* Have a smart phone (iPhone or Android device) with Wi-Fi internet connection at home.
* Actively using an email account
* Willing to accept the random study assignment.
* Willing to wear a Fitbit band 'a physical activity tracking device' on your wrist for five weeks every single day.
* Willing to have an Echo speaker 'a smart home speaker with voice assistant' installed in your home and use the digital voice assist for four weeks.
* Willing to receive daily text messages on your phone for four weeks.
* Willing to provide us with access to your Fitbit physical activities data.
* Willing to sign the consent form.

Exclusion Criteria:

* Already doing moderate to high physical activities in their daily life (rapid screener).
* Planning to relocate within the next 4-5 weeks.
* Stage 4 cancer.
* Already using physical activity tracker or part of a physical activity program.
* Part of another study that may interfere with our outcome of interest, unstable mental condition.
* Mental condition that prevents patient from performing the study activities and requirements.
* Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Average number of steps. Wearable sensor based | 5 weeks
  The investigators will measure your physical activity by number of steps before and after intervention via wearable activity tracker.

SECONDARY OUTCOMES:
Total number and duration of activity bouts. Wearable sensor based | 5 weeks
  Defined as 3 min. or more of uninterrupted activity measured by wearable sensor.
Transitions between active/inactive periods. Wearable sensor based | 5 weeks
  Time spent walking vs time spent sitting measured by all in one sensor.
Daily patterns of activity. Wearable sensor based | 5 weeks
  Distribution parameter of number of steps per/minute within 24 hours period. Measured by all in one sensor.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hassoon, MD,MPH,PMP, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hassoon A, Baig Y, Naiman DQ, Celentano DD, Lansey D, Stearns V, Coresh J, Schrack J, Martin SS, Yeh HC, Zeilberger H, Appel LJ. Randomized trial of two artificial intelligence coaching interventions to increase physical activity in cancer survivors. NPJ Digit Med. 2021 Dec 9;4(1):168. doi: 10.1038/s41746-021-00539-9. PMID 34887491
- [Derived] Hassoon A, Schrack J, Naiman D, Lansey D, Baig Y, Stearns V, Celentano D, Martin S, Appel L. Increasing Physical Activity Amongst Overweight and Obese Cancer Survivors Using an Alexa-Based Intelligent Agent for Patient Coaching: Protocol for the Physical Activity by Technology Help (PATH) Trial. JMIR Res Protoc. 2018 Feb 12;7(2):e27. doi: 10.2196/resprot.9096. PMID 29434016